CLINICAL TRIAL: NCT02314936
Title: Dose-ranging Efficacy of Supplementation With Polydextrose, a Dietary Fibre, on Colonic Transit Time and Gastrointestinal Symptoms in Adults With Functional Constipation: A Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Dose-ranging Efficacy of Polydextrose Supplement on Colonic Transit Time and Symptoms in Adults With Functional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: DuPont Nutrition and Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 01-2014
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-04

CONDITIONS: Functional Constipation
Keywords: Constipation; Polydextrose; Dietary Fiber; PAC-QoL; Colonic Transit Time; PAC-SYM
MeSH Terms: conditions — Constipation | interventions — polydextrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Litesse powder containing 12 g polydextrose (Experimental): 12 g of polydextrose, 1 sachet of powder mixed with water taken daily with breakfast for 2 weeks
  Interventions: Dietary Supplement: Litesse powder containing 12 g polydextrose
- Litesse powder containing 8 g polydextrose (Experimental): 8 g of polydextrose, 1 sachet of powder mixed with water taken daily with breakfast for 2 weeks
  Interventions: Dietary Supplement: Litesse powder containing 8 g polydextrose
- Litesse powder containing 4 g polydextrose (Experimental): 4 g of polydextrose, 1 sachet of powder mixed with water taken daily with breakfast for 2 weeks
  Interventions: Dietary Supplement: Litesse powder containing 4 g polydextrose
- Placebo (Placebo Comparator): Maltodextrin, 1 sachet of powder mixed with water taken daily with breakfast for 2 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Litesse powder containing 12 g polydextrose — 12 g polydextrose
  Other Names: Litesse powder
  Arms: Litesse powder containing 12 g polydextrose
Dietary Supplement: Litesse powder containing 8 g polydextrose — 8 g polydextrose, 4 g maltodextrin
  Other Names: Litesse powder
  Arms: Litesse powder containing 8 g polydextrose
Dietary Supplement: Litesse powder containing 4 g polydextrose — 4 g polydextrose, 8 g maltodextrin
  Other Names: Litesse powder
  Arms: Litesse powder containing 4 g polydextrose
Dietary Supplement: Placebo — 12 g Maltodextrin
  Arms: Placebo

SUMMARY:
This study will investigate the effectiveness of Polydextrose, a dietary fiber, at decreasing Colonic Transit Time and the gastrointestinal symptoms of Functional Constipation. One quarter of the subjects will receive 12 g of Polydextrose daily, one quarter will receive 8 g of Polydextrose daily, one quarter will receive 4 g of Polydextrose daily and one quarter will receive a placebo daily.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years.
2. Body mass index between 18.5 and 29.9 kg/m2 (encompasses normal weight and overweight).
3. If female, subject is not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation).

   OR

   Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:

   Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System), Intrauterine devices, Double barrier method, Vasectomy of partner (shown successful as per appropriate follow-up), Tubal ligation, and Non-heterosexual lifestyle (same sex partner).
4. Meets the Rome III criteria for functional constipation as follows: (Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis):

   Must meet 2 or more of the following criteria:

   Straining during at least 25% of defecations, Lumpy or hard stools in at least 25% of defecations, Sensation of incomplete evacuation for at least 25% of defecations, Sensation of anorectal obstruction/blockage for at least 25% of defecations, Manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor)

   Fewer than three defecations per week

   Loose stools are rarely present without the use of laxatives

   Insufficient criteria for irritable bowel syndrome
5. Ability of the participant (in the investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects.
6. Consent to the study and willing to comply with study product and methods.
7. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

1. Major gastrointestinal complication (e.g. Crohn's disease, colitis, celiac disease)
2. Prior abdominal surgery that in the opinion of the investigator may present a risk for the subject or confound study results.
3. Clinically significant underlying systemic illness that may preclude the participant's ability to complete the trial or that may confound the study outcomes (e.g. bowel cancer, prostate cancer, terminal illness).
4. Daily consumption of probiotics, prebiotics, fermented milk, and/or yogurt within 2 weeks of screening and throughout the trial other than the provided study products.
5. Laxative use within 48 hours of screening (rescue medication allowed for intolerable symptoms during study).
6. Regular use of any drug or dietary supplement known to cause constipation (e.g. iron, opioids, sucralfate, misoprostol, 5-HT#-antagonists, antacids with magnesium, calcium or aluminum, antidiarrheal medication, anticholinergic agents, calcium supplements, calcium channel blockers, tricyclic antidepressants or NSAIDs), within 1 month before screening.
7. Anticipated major dietary or exercise changes during the study.
8. Systemic steroid use, within 1 month before screening.
9. Eating disorder.
10. Contraindication to dairy products (e.g., intolerance to lactose or any substance in the study product).
11. History of alcohol, drug, or medication abuse.
12. Pregnant or lactating female, or pregnancy planned during study period.
13. Participation in another study with any investigational product within 60 days of screening.
14. Investigator believes that the participant may be uncooperative and/or noncompliant and should therefore not participate in the study.
15. Subject under administrative or legal supervision.
16. Subject who would receive more than 4500 Euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Started | 48 | 48 | 48 | 48
Completed | 48 | 48 | 46 | 48
Not Completed | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo | Total
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (16.3) | 42.9 (12.5) | 41.5 (17.1) | 43.6 (13.4) | 42.7 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 32 | 33 | 133
  Male | 14 | 14 | 16 | 15 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 0 | 0 | 0 | 2
  Central American | 2 | 1 | 0 | 1 | 4
  East Asian | 1 | 0 | 1 | 2 | 4
  Eastern European White | 0 | 3 | 0 | 5 | 8
  Middle Eastern | 2 | 1 | 2 | 1 | 6
  North American Indian | 0 | 0 | 2 | 0 | 2
  South American | 0 | 6 | 3 | 3 | 12
  South Asian | 3 | 1 | 0 | 1 | 5
  South East Asian | 2 | 0 | 0 | 0 | 2
  Western European White | 36 | 36 | 40 | 35 | 147
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.27 (3.06) | 25.31 (3.09) | 25.32 (2.82) | 25.23 (2.48) | 25.28 (2.85)
Smoking Status [Count of Participants; unit: Participants]
  Ex-Smoker | 7 | 8 | 3 | 7 | 25
  Non-Smoker | 34 | 36 | 40 | 35 | 145
  Current Smoker | 7 | 4 | 5 | 6 | 22
Alcohol Use [Count of Participants; unit: Participants]
  Daily | 0 | 2 | 2 | 1 | 5
  None | 9 | 5 | 9 | 9 | 32
  Occasionally | 27 | 25 | 21 | 27 | 100
  Weekly | 12 | 16 | 16 | 11 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change in Colonic Transit Time From Baseline to Day 15
Description: Assessed using abdominal x-ray. Subjects will take 24 radiopaque markers for 6 consecutive days (144 radiopaque markers in total) immediately preceding the x-ray dates.
Time Frame: Baseline and Day 15
Population: The number of participants analysed is the number of participants who met the per protocol population requirement. 17 participants did not meet the per protocol compliance (must have consumed ≥80% of assigned study product and 100% of radio opaque pellets) and 2 participants did not complete the study (did not complete end-of-study visit).
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
Hours | -1.7 (23.6) | 4.0 (23.4) | 2.5 (23.7) | 2.6 (25.9)

2. Secondary Outcome: Change in Participant Assessment of Constipation Symptoms (PAC-SYM) From Baseline to Day 15
Description: Assessed using the PAC-SYM questionnaire (overall score, abdominal symptoms score, rectal symptoms score, and stool symptoms score).
  The PAC-SYM was developed as a brief, easily administered tool to assess symptom frequency and severity of chronic constipation. The authors used a definition for constipation was based on the Rome II criteria. This 12-item self-report measure is divided into the 3 symptom subscales of: abdominal, rectal and stool subscales.
  All items (sub-scores and the total score) are scored on a five-point Likert scale ranging from 0 (absence of symptom) to 4 (very severe) where lower scores are better. Scores for the total number of non-missing items within the subscale or total score are summed and divided by the total number of non-missing items for that subscale or total score.
Time Frame: Baseline and Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
scores on a scale
  Overall Score | -0.24 (0.59) | -0.13 (0.39) | -0.04 (0.44) | -0.21 (0.56)
  Abdominal Symptoms Score | -0.13 (0.69) | -0.06 (0.51) | -0.01 (0.56) | -0.15 (0.60)
  Rectal Symptoms Score | -0.28 (0.71) | -0.16 (0.46) | 0.06 (0.60) | -0.21 (0.59)
  Stool Symptoms Score | -0.31 (0.82) | -0.16 (0.68) | -0.18 (0.62) | -0.28 (0.82)

3. Secondary Outcome: Change in Participant Assessment of Constipation Quality of Life (PAC-QoL) From Baseline to Day 15
Description: Assessed using the PAC-QoL questionnaire (Overall Score, Worries and Concerns Score, Physical Discomfort Score, Psychosocial Discomfort Score, and Satisfaction Score)
  The Patient Assessment of Constipation (PAC) was developed to address the need for a disease-specific patient-reported outcomes measure. It includes components from complementary symptom and quality of life questionnaires.
  The PAC-QOL contains 28 items grouped into 4 subscales covering: worries and concerns (11 items), physical discomfort (4 items), psychosocial discomfort (8 items), and satisfaction (5 items).
  A 5-point Likert response scale, ranging from 0 (not at all / none of the time) to 4 (extremely / all of the time), where lower scores are better. Scores are computed as the average non-missing item response within the subscale where each score is given equal weight; the global score is calculated as the mean of the 28-items.
Time Frame: Baseline and Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
scores on a scale
  Overall Score | -0.05 (0.36) | -0.04 (0.45) | -0.08 (0.33) | -0.11 (0.33)
  Worries and Concerns Score | -0.27 (0.59) | -0.17 (0.54) | -0.15 (0.46) | -0.13 (0.60)
  Physical Discomfort Score | -0.24 (0.74) | -0.23 (0.73) | -0.13 (0.58) | -0.20 (0.75)
  Psychosocial Discomfort Score | -0.12 (0.53) | -0.11 (0.58) | -0.17 (0.52) | -0.09 (0.53)
  Satisfaction Score | 0.44 (0.98) | 0.37 (0.75) | 0.12 (0.67) | -0.02 (0.69)

4. Secondary Outcome: Change in Bowel Function Index From Baseline to Day 15
Description: Assessed using the Bowel Function Index questionnaire (total score, ease of defecation, feeling of incomplete bowel evacuation, and personal judgement of constipation).
  Each of the three questions used a numerical analog scale (0 = easy/no difficulty/not at all, 100 = very strong/very difficult) for grading purposes. The three questions were calculated as single scores as well as by a total score defined as the average of the three questions.
Time Frame: Baseline and Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
scores on a scale
  Overall Score | -9.3 (23.6) | -8.2 (20.8) | -8.9 (20.1) | -10.2 (23.4)
  Ease of Defecation | -6.2 (32.8) | -6.2 (26.1) | -5.9 (26.2) | -8.8 (25.8)
  Feeling of Incomplete Bowel Evacuation | -11.6 (30.1) | -10.9 (31.5) | -15.1 (23.3) | -9.5 (34.0)
  Personal Judgement of Constipation | -10.1 (27.3) | -7.5 (24.3) | -5.7 (20.9) | -12.4 (27.6)

5. Secondary Outcome: Change in Adequate Relief of Constipation Symptoms From Baseline to Day 15
Description: Assessed using single question dichotomous tool.
  Adequate relief quantified the difference in the number of participants experiencing relief from constipation between participants supplemented with Litesse and those supplemented with a placebo at baseline and day 14. The units of analysis for the relief questionnaire were the number of participants who reported relief from constipation.
Time Frame: Baseline and Day 15
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
Participants
  Relief at Baseline | 24 | 25 | 19 | 16
  Relief at Day 14 End-of-Study | 36 | 31 | 20 | 26

6. Secondary Outcome: Change in Stool Frequency From Baseline to Day 15
Description: Participants will record the number of defecations per day in a daily diary
Time Frame: 14 day run-in and Week 2 of the 14-day supplementation period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Bowel Movements Per Day
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
Number of Bowel Movements Per Day | 1.2 (3.3) | -0.2 (3.3) | -0.4 (2.2) | -0.9 (3.7)

7. Secondary Outcome: Change in Stool Consistency From Baseline to Day 15
Description: Stool consistency will be rated each day in a diary by using the Bristol Stool Scale Form.
  Bristol Stool Scale:
  The BSS is a categorical scale ranging from 1 to 7 that interprets the consistency of a single bowel movement; a single score is recorded and used for analysis. Lower scores are associated with hard and lumpy consistencies while higher scores are associated with soft or liquid consistencies. Generally, an optimal BSS scores ranges from 3 to 5.
Time Frame: 14 day run-in and Week 2 of the 14-day supplementation period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
scores on a scale | 0.33 (0.99) | -0.11 (0.95) | 0.30 (0.99) | 0.13 (0.93)

8. Secondary Outcome: Change in the Degree of Straining During Defecation From Baseline to Day 15
Description: Degree of straining for each bowel movement will be recorded in a daily diary using a 5-point scale.
  The degree of straining is a rating scale ranging from 1 (not at al) to 5 (an extreme amount) that interprets the degree to which an individual must strain during a unique defecation; a single core is recorded and used for analysis. Scores were calculated as the weekly average of the daily degree of straining (1-5) where a lower score represented less straining.
Time Frame: 14 day run-in and Week 2 of the 14-day supplementation period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
scores on a scale | -0.07 (0.82) | -0.26 (0.87) | -0.15 (0.81) | -0.09 (0.46)

9. Secondary Outcome: Change in the Sensation of Complete Bowel Emptying From Baseline to Day 15
Description: Sensation of complete bowel emptying for each bowel movement will be recorded in a daily diary on a dichotomous "yes" or "no" scale.
  The change in the sensation was defined as the change from baseline to week 2 in the percentage of complete bowel movements (CBMs) between participants supplemented with Litesse and those supplemented with a placebo. It assessed whether the participant felt as though their bowel movement was complete. The units of analysis for the sensation of complete bowel emptying was the weekly percentage of complete bowel movements, for each participant at run-in (week -1), week 1 and week 2.
Time Frame: 14 day run-in and Week 2 of the 14-day supplementation period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of CBMs per week
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
Percentage of CBMs per week | 10.8 (27.5) | 10.2 (25.1) | 7.3 (31.3) | -3.4 (33.2)

10. Secondary Outcome: Change in the Severity of Abdominal Discomfort From Baseline to Day 15
Description: Severity of abdominal discomfort will be recorded each day in a daily diary on a 5-point scale.
  The severity of abdominal discomfort was calculated from a rating scale ranging from 1 (not at all) to 5 very severe); a single score was recorded and used for analysis. Scores were calculated as the weekly average of the daily degree of discomfort where a lower score represented less straining.
Time Frame: 14 day run-in and Week 2 of the 14-day supplementation period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
scores on a scale | 0.06 (0.57) | -0.05 (0.61) | -0.10 (0.58) | -0.01 (0.44)

11. Secondary Outcome: Change in the Bloating Severity From Baseline to Day 15
Description: Severity of bloating will be recorded each day in a daily diary on a 5-point scale.
  The severity of abdominal bloating was calculated from a rating scale ranging from 1 (not at all) to 5 very severe); a single score was recorded and used for analysis. Scores were calculated as the weekly average of the daily degree of bloating where a lower score represented less straining.
Time Frame: 14 day run-in and Week 2 of the 14-day supplementation period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
scores on a scale | -0.13 (0.58) | -0.23 (0.47) | -0.12 (0.49) | -0.03 (0.58)

12. Secondary Outcome: Overall Product Satisfaction
Description: Participants will be asked to rate their overall satisfaction with the study product's ability to relieve their constipation symptoms on a 5-point ordinal scale.
  The overall product satisfaction questionnaire consists of a single question that provides insight regarding the participants satisfaction on the product's ability to relieve constipation symptoms. The score that the participant indicates is considered the total score and no sub-scores are calculated. It is a rating scale that ranges from 1 (not at all satisfied) to 5 (very satisfied) where a higher score at the end-of-study indicates an improvement.
Time Frame: Assessed at Day 15 (end of study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
scores on a scale | 3.26 (1.20) | 3.09 (1.23) | 2.54 (1.14) | 2.62 (1.15)

13. Other Pre Specified Outcome: Change in Hemoglobin Levels From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically hemoglobin in this outcome).
Time Frame: Screening and Day 15 (end of study)
Population: Whole blood hematology was not obtained from two participants (one participant in the Litesse powder containing 12 g polydextrose arm and one participant in the Litesse powder containing 4 g polydextrose).
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
g/dL | -1.0 (5.1) | -0.9 (5.5) | -1.4 (5.1) | 0.3 (5.7)

14. Other Pre Specified Outcome: Change in Hematocrit Levels From Screening to Day 15
Description: Safety will be evaluated by measuring the change in whole blood hematology (specifically hematocrit levels in this outcome).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
Percentage of red blood cells | -0.0045 (0.0156) | -0.0008 (0.0166) | -0.0057 (0.0141) | 0.0031 (0.0146)

15. Other Pre Specified Outcome: Change in White Blood Cell Count From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically white blood cell count in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
10^9 cells/L | 0.13 (1.56) | -0.34 (1.19) | -0.19 (1.24) | 0.06 (1.33)

16. Other Pre Specified Outcome: Change in Red Blood Cell Count From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically red blood cell count in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
10^12 cells/L | -0.052 (0.157) | -0.030 (0.171) | -0.053 (0.163) | 0.034 (0.159)

17. Other Pre Specified Outcome: Change in Mean Corpuscular Volume From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically mean corpuscular volume in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
fL | 0.10 (1.13) | 0.23 (1.09) | -0.19 (1.21) | -0.09 (1.05)

18. Other Pre Specified Outcome: Change in Mean Corpuscular Hemoglobin From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically mean corpuscular hemoglobin in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
pg | 0.16 (0.75) | -0.02 (0.63) | 0.04 (0.46) | -0.15 (0.54)

19. Other Pre Specified Outcome: Change in Mean Corpuscular Hemoglobin Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically mean corpuscular hemoglobin concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
g/dL | 0.8 (5.2) | -0.9 (5.9) | 1.4 (4.7) | -1.5 (5.5)

20. Other Pre Specified Outcome: Change in Red Cell Distribution Width From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically red cell distribution width in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent of mean red blood cell volume
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
percent of mean red blood cell volume | -0.03 (0.35) | 0.06 (0.33) | -0.03 (0.62) | -0.08 (0.43)

21. Other Pre Specified Outcome: Change in Platelet Count From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically platelet count in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
10^9 cells/L | -3.7 (20.4) | 6.0 (27.0) | -5.9 (25.9) | 1.6 (29.5)

22. Other Pre Specified Outcome: Change in Neutrophil Count From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically neutrophil count in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
10^9 cells/L | 0.10 (1.43) | -0.19 (1.00) | -0.19 (1.00) | 0.10 (1.05)

23. Other Pre Specified Outcome: Change in Lymphocyte Count From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically lymphocyte count in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
10^9 cells/L | 0.04 (0.44) | -0.10 (0.36) | -0.01 (0.39) | -0.06 (0.48)

24. Other Pre Specified Outcome: Change in Monocyte Count From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically monocyte count in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
10^9 cells/L | -0.002 (0.39) | -0.012 (0.13) | -0.006 (0.139) | 0.021 (0.160)

25. Other Pre Specified Outcome: Change in Eosinophil Count From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically eosinophil count in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
10^9 cells/L | -0.002 (0.090) | -0.025 (0.076) | 0.030 (0.197) | 0.029 (0.153)

26. Other Pre Specified Outcome: Change in Basophil Count From Baseline to Day 15
Description: Safety will be evaluated by measuring whole blood hematology (specifically basophil count in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 48 | 47 | 48
10^9 cells/L | 0.000 (0.042) | 0.008 (0.050) | 0.002 (0.033) | 0.010 (0.037)

27. Other Pre Specified Outcome: Change in Serum Glucose Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically glucose concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: The number analyzed from the Litesse powder 4g arm is only 47 due to laboratory analysis error.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 48
mmol/L | -0.12 (0.42) | 0.04 (0.46) | -0.15 (0.44) | -0.10 (0.57)

28. Other Pre Specified Outcome: Change in Creatinine Levels in Blood From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically creatinine concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: μmol
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
μmol | 0.8 (8.4) | -0.1 (5.9) | 0.6 (4.8) | 0.8 (5.4)

29. Other Pre Specified Outcome: Change in Serum Urea Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically urea concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
mmol/L | 0.18 (1.11) | -0.31 (1.00) | -0.10 (1.03) | 0.08 (1.20)

30. Other Pre Specified Outcome: Change in Serum Estimated Globular Filtration Rate From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically estimated glomerular filtration rate in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
mL/min/1.73m^2 | -1.9 (10.8) | 1.4 (7.8) | -0.1 (5.6) | -1.9 (6.3)

31. Other Pre Specified Outcome: Change in Serum Sodium Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically sodium concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
mmol/L | -0.90 (2.94) | -0.27 (2.30) | -0.83 (2.60) | -0.19 (2.50)

32. Other Pre Specified Outcome: Change in Serum Potassium Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically potassium concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: One participant in the Litesse powder containing 4 g polydextrose arm did not have this blood serum variable analysed due to laboratory analysis error.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 48
mmol/L | -0.21 (0.53) | -0.01 (0.61) | -0.21 (0.50) | -0.01 (0.46)

33. Other Pre Specified Outcome: Change in Serum Chloride Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically chloride concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
mmol/L | -0.21 (2.32) | -0.004 (2.40) | -0.71 (2.08) | -0.29 (2.28)

34. Other Pre Specified Outcome: Change in Serum Calcium Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically calcium concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
mmol/L | -0.019 (0.101) | 0.016 (0.092) | -0.004 (0.085) | 0.028 (0.098)

35. Other Pre Specified Outcome: Change in Serum Carbon Dioxide Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically carbon dioxide concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 48
mmol/L | -0.60 (2.73) | 0.31 (2.49) | -0.13 (2.65) | -0.50 (2.26)

36. Other Pre Specified Outcome: Change in Serum Phosphate Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically phosphate concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
mmol/L | 0.011 (0.147) | -0.034 (0.165) | 0.012 (0.168) | -0.003 (0.244)

37. Other Pre Specified Outcome: Change in Serum Bilirubin Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically bilirubin concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
μmol/L | -0.5 (4.0) | 0.6 (3.3) | 0.1 (3.4) | 0.6 (5.0)

38. Other Pre Specified Outcome: Change in Serum Aspartate Transaminase Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically aspartate transaminase concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
U/L | 0.7 (4.5) | 3.2 (16.2) | -0.1 (7.8) | 0.2 (4.9)

39. Other Pre Specified Outcome: Change in Serum Alanine Transaminase Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically alanine transaminase concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
U/L | 1.6 (7.0) | -0.1 (7.7) | -1.0 (9.5) | -0.6 (8.2)

40. Other Pre Specified Outcome: Change in Serum Alkaline Phosphate Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically alkaline phosphate concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
U/L | 1.0 (6.7) | -0.7 (7.7) | -1.0 (7.0) | 1.9 (9.8)

41. Other Pre Specified Outcome: Change in Serum Gamma-Glutamyltransferase Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically gamma-glutamyltransferase concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
U/L | 0.6 (4.0) | -1.6 (6.1) | 0.3 (6.2) | -2.8 (15.3)

42. Other Pre Specified Outcome: Change in Serum C-Reactive Protein Concentration From Baseline to Day 15
Description: Safety will be evaluated by measuring blood serum variables (specifically C-reactive protein concentration in this outcome measure).
Time Frame: Screening and Day 15 (end of study)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
mg/L | 0.6 (2.6) | 0.1 (4.4) | -0.2 (2.4) | 0.4 (2.6)

43. Other Pre Specified Outcome: Change in Specific Gravity Urinalysis Parameter From Screening to Day 15
Description: Safety will be evaluated by measuring urine analyses (specifically specific gravity in this outcome measure). The reference range for specific gravity are 1.001 - 1.030 mmol/L, with no alerting or critical values.
Time Frame: Screening and Day 15 (end of study)
Population: One participant from the 12 g polydextrose arm, one participant from the 8 g polydextrose arm, and three participants from the 4 g polydextrose arm were unable to have urinalysis parameters analysed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 47 | 45 | 48
mmol/L | 0.0010 (0.0072) | 0.0007 (0.0071) | 0.0005 (0.0135) | 0.0029 (0.0096)

44. Other Pre Specified Outcome: Change in pH Urinalysis Parameter From Baseline to Day 15
Description: Safety will be evaluated by measuring urine analyses (specifically urine pH in this outcome measure). Urine pH reference range is between 5.0 - 8.0, with no alerting or critical values.
Time Frame: Screening and Day 15 (end of study)
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 47 | 47 | 45 | 48
pH | -0.05 (0.97) | 0.20 (1.10) | 0.02 (1.02) | 0.06 (1.07)

45. Other Pre Specified Outcome: Number of Subjects With Adverse Events
Description: Adverse events were recorded in a daily diary during the 14-day run-in period and the 14-day treatment period. All types of adverse events as well as the total number of all adverse events reported were used in this outcome measure.
Time Frame: 14 days run-in and 14 days treatment
Population: as for outcome 1
Measure: Number; unit: Number of Adverse Events
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Number analyzed (Participants) | 45 | 43 | 43 | 42
Number of Adverse Events | 30 | 23 | 11 | 29

ADVERSE EVENTS:
Time Frame: Adverse events were reported between Day -14 to Day 14 (run-in and intervention periods).
Arm/Group | Litesse Powder Containing 12 g Polydextrose | Litesse Powder Containing 8 g Polydextrose | Litesse Powder Containing 4 g Polydextrose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 11/48 | 10/48 | 1/48 | 11/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Litesse Powder Containing 12 g Polydextrose (N=48) | Litesse Powder Containing 8 g Polydextrose (N=48) | Litesse Powder Containing 4 g Polydextrose (N=48) | Placebo (N=48)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (3)
Abdominal Distension (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 3 (3)
Frequent Bowel Movements (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 0 (0) | 4 (4)

LIMITATIONS AND CAVEATS:
The study population was not sufficiently constipated at baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes